CLINICAL TRIAL: NCT01868191
Title: Effects of Benfotiamine on Intraepidermal Nerve Fiber Density (IENFD)and Diabetic Neuropathy in Subjects With Sensorimotor Diabetic Polyneuropathy: a Double-blind, Randomized, Placebo-controlled Parallel Group Pilot Study Over 12 Months.
Brief Title: Effects of Benfotiamine on Intraepidermal Nerve Fiber Density (IENFD)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diabetes Schwerpunktpraxis (Other)
Collaborators: Woerwag Pharma GmbH & Co. KG (Industry)
Responsible Party: Principal Investigator, Ovidiu Alin Stirban, Dr. med., Diabetes Schwerpunktpraxis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WOE_2013_SB
Record Dates: First submitted 2013-05-25; First posted 2013-06-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetes; Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus | interventions — benphothiamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo for benfotiamine (Placebo Comparator): Placebo for benfotiamine 600 mg/day for the first 3 months followed by 300 mg/day for 9 months
  Interventions: Drug: Placebo for benfotiamine
- Benfotiamine (Experimental): Treatment with benfotiamine 600 mg/day for 3 months followed by 300 mg/day for 9 months
  Interventions: Drug: Benfotiamine

INTERVENTIONS:
Drug: Benfotiamine — Treatment with 600 mg/day for the first 3 months followed by 300 mg/day for 9 months
  Other Names: Milgamma protekt
  Arms: Benfotiamine
Drug: Placebo for benfotiamine — Treatment with placebo for benfotiamine 600 mg/day for the first 3 months followed by 300 mg/day for 9 months
  Arms: Placebo for benfotiamine

SUMMARY:
The aim of the present study is to assess before, as well as 6 and 12 months following a therapy with benfotiamine the influence of therapy on intraepidermal nerve fiber density (skin biopsy) and neuropathic symptoms and deficits in people with type 1 or 2 diabetes mellitus and diabetic sensomotoric neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Have type 1 or type 2 diabetes mellitus based on the disease diagnostic criteria (WHO) classification on ongoing insulin or/and oral antidiabetic therapy with a stable regimen for the previous 3 months
* Male or female subjects aged between 18 and 75 years, inclusive
* Have an HbA1c level ≤ 9.5% without optimizing potential
* mTCNS (modified Toronto Clinical Neuropathy Score) ≥ (above or equal to) 6) OR (a score on the MNSI (Michigan Neuropathy Screening Instrument)questionnaire of ≥4 or a score on the MNSI examination ≥2.5)
* Medical history without major pathology (with the exception of type 2 diabetes) as judged by the investigator, especially no major peripheral artery disease.
* Body mass index (BMI) between 25 and 45kg/m2, both inclusive

Exclusion Criteria:

* Subjects with secondary forms of diabetes such as due to pancreatitis.
* Current or previous treatment (less than 6 months) with benfotiamine, B-vitamins, vitamin B complex, alpha lipoic acid or actovegin.
* Have any contraindications, known allergy, or hypersensitivity to benfotiamine.
* Have any contraindications, known allergy, or hypersensitivity to local anesthetics.
* Neuropathy by other origin than diabetes.
* Other severe pain that might impair the assessment of neuropathic pain.
* Treatment with more than one of following: tricyclic antidepressants, serotonin norepinephrine reuptake inhibitors, anticonvulsants, class I antiarrhythmics with Na-channel inhibition (mexiletine, flecainid, propafenon and others) or neuroleptics in patients receiving these drugs for neuropathic pain.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in intraepidermal nerve fiber density | 6 and 12 months

SECONDARY OUTCOMES:
Change in neuropathic symptoms | 3, 6 and 12 months
  Following questionnaires will be used to assess neuropathic symptoms: modified Toronto Clinical Neuropathy Score and Michigan Neuropathy Screening Instrument
Change in neuropathic deficits | 3, 6 and 12 months
  A score will be calculated at each timepoint using the Michigan Neuropathy Screening Instrument

CONTACTS AND LOCATIONS:
Overall Officials: Alin O Stirban, MD, PhD, Principal Investigator — Diabetes Schwerpunktpraxis
Locations (1):
- Diabetes Schwerpunktpraxis, Essen, North Rhine-Westphalia, Germany